CLINICAL TRIAL: NCT01770626
Title: A Pilot Study to Determine the Effectiveness of Bioelectrical Impedance Analysis as a Clinical Assessment Tool of Nutrition Status in Glioblastoma Multiforme Patients (The BEAM Study [BIA Effectiveness as Assessment Tool for Glioblastoma Multiforme (GBM) Patients])
Brief Title: A Pilot Study to Determine Nutrition Status in Glioblastoma Multiforme Patients
Acronym: BEAM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UAB 1106
Record Dates: First submitted 2012-12-20; First posted 2013-01-18 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Brain Cancer
MeSH Terms: conditions — Brain Neoplasms | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (No Intervention): evaluate the composition of a participant's body, diagnosed with a brain tumor (glioblastoma multiforme) as determined by bioelectrical impedance analysis
  Interventions: Other: Nutrition

INTERVENTIONS:
Other: Nutrition — Anthropometrics, Nutrition assessment, Bioelectrical Impedance Analysis, Blood sample, Resting Energy Expenditure. All will be done 2-3 weeks after initial study visit and will continue every 3 months study visit except the Resting Energy Expenditure which will be performed at only one visit (2-3 weeks after initial visit).

SUMMARY:
The study is designed to evaluate how the composition of a participant's body, diagnosed with a brain tumor (glioblastoma multiforme) as determined by bioelectrical impedance analysis can predict the progression and outcomes of disease.

DETAILED DESCRIPTION:
The purpose of this study is to monitor the nutritional status of (Glioblastoma Multiforme)GBM patients for one year. We will look at the relationships between phase angle determined by Bioelectrical Impedance Analysis (BIA), nutrition assessment by Subjective Global Assessment and serum albumin, the type of microbes present in the gut, the participant's DNA information, and tumor progression. We will also compare estimated caloric needs determined by BIA and Harris Benedict Equation to Resting Energy Expenditure from Indirect Calorimetry of the people with GBM and the people without.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 19 years of age.
* Subjects must have a histologically confirmed supratentorial grade IV astrocytoma (glioblastoma multiforme).
* Women of childbearing potential must have a negative pregnancy test.

Exclusion Criteria:

* Subjects with implanted pacemakers or defibrillators.
* Subjects who are pregnant.
* Subjects with edema.
* Subjects with an amputated extremity.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-07 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the use of Bioelectrical Impedance Analysis as a clinical assessment tool in Glioblastoma Multiforme patients | Participants will be followed every 3 months up to 12 months
  The electrical current used by the BIA (Bioelectrical Impedance Analysis) is low and below the level. The electrodes will be placed on hand and foot.

SECONDARY OUTCOMES:
To compare estimated caloric needs determined by BIA and Harris Benedict Equation to Resting Energy Expenditure from Indirect Calorimetry | At initial visit until end of study.Participants will be followed for duration average of every 3 months
  Age, sex, and body composition are the prime influences on resting energy expenditure (REE), the energy used by an individual when fasted and at rest. The largest component of total energy expenditure (TEE) is REE.

CONTACTS AND LOCATIONS:
Overall Officials: Louis B Nabors, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States